CLINICAL TRIAL: NCT06324305
Title: Comparative Study Between Three Different Techniques in Drainage of Sub-Retinal Fluid During Pars Plana Vitrectomy for Patients With Macula Off Rhegmatogenous Retinal Detachment
Brief Title: Comparative Study Between Three Different Techniques in Drainage of SRF During PPV in RRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina tarek mohamed kamel, Dina kamel, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRF drainage techniques in RRD
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: drainage techniquies; comparison; subretinal fluid
MeSH Terms: interventions — Predictive Value of Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): drainage of sub-retinal fluid from the original (primary) break
  Interventions: Procedure: Pars plana vitrectomy (PPV) and drainage of subretinal fluid
- Group 2 (Active Comparator): drainage of sub-retinal fluid using perfluorocarbon (PFC) and removing sub-retinal fluid through the original break or peripheral retinotomy
  Interventions: Procedure: Pars plana vitrectomy (PPV) and drainage of subretinal fluid
- Group 3 (Active Comparator): drainage of sub-retinal fluid through formation of a posterior drainage retinotomy only.
  Interventions: Procedure: Pars plana vitrectomy (PPV) and drainage of subretinal fluid

INTERVENTIONS:
Procedure: Pars plana vitrectomy (PPV) and drainage of subretinal fluid — Drainage of subretinal fluid during Pars Plana Vitrectomy in patients with rhegmatogenous retinal detachment (RRD)

SUMMARY:
The study will investigate and compare the three techniques in drainage of subretinal fluid in patients with macula off RRD: namely using the original break, performing a posterior drainage retinotomy and using PFC with drainage through the original break or peripheral retinotomy regarding the presence of persistent sub-retnal fluid and related intra or postoperative complications

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment (RRD) is a serious surgical condition with significant ocular morbidity if not managed properly. Approaches to the repair of RRD have greatly evolved over the years, leading to outstanding primary surgical success rates. The management of RRD is often a topic of great debate. Several factors may affect surgical success and dictate a surgeon's preference for the technique employed.

Scleral buckling, vitrectomy and pneumatic retinopexy have been used successfully for the treatment of RRD.

Using original breaks to drain subretinal fluid without perfluorocarbon liquid in cases of vitrectomy for RRD may be an effective and safe surgical technique for functional and anatomical recovery without serious complications. but it may leave some SRF at the macula (2) Posterior drainage retinotomy is a surgical technique that involves the creation of a small retinal hole to facilitate the removal of subretinal fluid (SRF), in conjunction with pars plana vitrectomy (PPV), for the treatment of rhegmatogenous retinal detachment (RRD) (3). First described by Machemer in 1981 as a technique for relaxing the retina in proliferative vitreoretinopathy (PVR) and trauma (4), retinotomy has since expanded to include more indications for its use (5). In addition, the use of drainage retinotomy aids the management of bullous RRD, because the complete drainage of fluid significantly decreases the likelihood of retinal fold formation (6). Although there are benefits with retinotomy, complications associated with its use include visual field scotomas and PVR at the endodrainage retinotomy sites .

Perfluorocarbon liquid (PFC) has been a major milestone in vitrectomy surgery and is an invaluable tool in the repair of giant retinal tear-associated detachments (8). By stabilizing the mobile, detached retina, PFC reduces the risk of iatrogenic breaks, especially towards the periphery. PFC may also be useful to assist with subretinal fluid drainage in cases when the retinal break is anterior in order to avoid the need for a posterior drainage retinotomy.

Subretinal fluid that persists after pars plana vitrectomy for RRD is defined by being persistent for more than one month. While mostly benign, SRF has been shown to exhibit complications. Those include the development of macular hole (MH), permanent disruption of the outer retinal layers, subretinal fibrosis, macular edema, and epiretinal membranes affecting the visual outcome.

To the best of our knowledge, very limited reports studied the comparison between the three techniques in an anatomical along with a functional way, presence of subretinal fluid that persists after (PPV) for macula off RRD, or related intra and postoperative complications and also relating them to the functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* • Age: above 18 years old

  * Patients with rhegmatogenous retinal detachment (RRD) where the detachment is involving the macula.
  * Patients with proliferative vitreoretinopathy (PVR) no more than PVR -B.
  * Patients with peripheral break.
  * Duration of detachment: within one month.

Exclusion Criteria:

* • Patients with macula on RRD.

  * Patients with tractional retinal detachment.
  * Patients with giant retinal tear.
  * Patients with proliferative vitreoretinopathy (PVR) more than PVR -B.
  * More than one month duration of detachment.
  * Patients with posterior staphyloma.
  * Patients with recurrent retinal detachment.
  * Patients with full thickness macular hole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The presence versus absence of sub-macular fluid using each of the three different techniques in pars plana vitrectomy (PPV) | within 1 week and within 1 month from the PPV
  optical coherence tomography (OCT) imaging after PPV

CONTACTS AND LOCATIONS:
Overall Officials: Dina T Mohamed, master's, Principal Investigator — AinShams University; Tamer F Elewa, MD, Study Chair — AinShams University

REFERENCES:
- [Background] Warren A, Wang DW, Lim JI. Rhegmatogenous retinal detachment surgery: A review. Clin Exp Ophthalmol. 2023 Apr;51(3):271-279. doi: 10.1111/ceo.14205. Epub 2023 Jan 25. PMID 36640144
- [Background] Fu Y, Chen S, Gu ZH, Zhang YL, Li LY, Yang N. Natural history of persistent subretinal fluid following the successful repair of rhegmatogenous retinal detachment. Int J Ophthalmol. 2020 Oct 18;13(10):1621-1628. doi: 10.18240/ijo.2020.10.17. eCollection 2020. PMID 33078114
- [Background] Mimouni M, Jaouni T, Ben-Yair M, Almus S, Derman L, Ehrenberg S, Almeida D, Barak Y, Zayit-Soudry S, Averbukh E. PERSISTENT LOCULATED SUBRETINAL FLUID AFTER RHEGMATOGENOUS RETINAL DETACHMENT SURGERY. Retina. 2020 Jun;40(6):1153-1159. doi: 10.1097/IAE.0000000000002565. PMID 31241497
- [Background] Chen X, Zhang Y, Yan Y, Hong L, Zhu L, Deng J, Din Q, Huang Z, Zhou H. COMPLETE SUBRETINAL FLUID DRAINAGE IS NOT NECESSARY DURING VITRECTOMY SURGERY FOR MACULA-OFF RHEGMATOGENOUS RETINAL DETACHMENT WITH PERIPHERAL BREAKS: A Prospective, Nonrandomized Comparative Interventional Study. Retina. 2017 Mar;37(3):487-493. doi: 10.1097/IAE.0000000000001180. PMID 27429377